CLINICAL TRIAL: NCT01780649
Title: Evaluation of the Efficiency and Indications of IMSI in Comparison With ICSI in Case of Male Infertility
Brief Title: Evaluation of IMSI to Treat Male Infertility
Acronym: PHRC-IMSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08 117 01; Ministry of Health, PHRC N (Other Grant/Funding Number: Ministry of Health)
Record Dates: First submitted 2013-01-23; First posted 2013-01-31 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2013-01

CONDITIONS: Infertility
Keywords: IMSI; ICSI; ART Assisted reproductive technology; Spermatozoa; male infertility; vacuoles
MeSH Terms: conditions — Infertility; Infertility, Male | interventions — Sperm Injections, Intracytoplasmic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IMSI (Experimental): Intracytoplasmic Morphologically Selected Sperm Injection (IMSI)
  Interventions: Procedure: IMSI
- ICSI (Active Comparator): Intracytoplasmic sperm injection (ICSI)
  Interventions: Procedure: ICSI

INTERVENTIONS:
Procedure: IMSI — Intracytoplasmic Morphologically Selected Sperm Injection (IMSI) is a modification of IntraCytoplasmic Sperm Injection (ICSI) with a choice of the spermatozoon to be injected done at a 6000x magnification instead of 400x commonly used in ICSI
  Arms: IMSI
Procedure: ICSI — ICSI is largely choice of the spermatozoon to be injected done at a 400x magnification
  Other Names: Intracytoplasmic sperm injection (ICSI)
  Arms: ICSI

SUMMARY:
Intracytoplasmic Morphologically Selected Sperm (IMSI) is a modification of IntraCytoplasmic Sperm Injection (ICSI) with a choice of the spermatozoon to be injected done at a 6000x magnification instead of 400x commonly used in ICSI. The purpose of this study is to evaluate the efficiency and the indications of IMSI through a multicentric randomised trial.

DETAILED DESCRIPTION:
Intracytoplasmic sperm injection (ICSI) is largely used to treat male infertility. Usually, choice of the spermatozoon to be injected is done at a 400x magnification. Recently, a new microscopic technic (Intracytoplasmic Morphologically Selected Sperm Injection-IMSI) allows to make this choice at a 6000x magnification, which permits to identify sperm abnormalities such as nuclear vacuoles not seen in conventional ICSI. This selection may improve ICSI outcome. However only few data from randomised trials, have been published and the indications of IMSI remain to be identified. The present study aims to evaluate the efficiency and the indications of IMSI through a multicentric randomised trial. The patients enrolled in the study must present a male infertility and will have complete sperm examination, including morphology, DNA fragmentation and nuclear immaturity. The main endpoint will be the percentage of delivery.

ELIGIBILITY:
Inclusion Criteria:

* male infertility with less than 1 million of motile spermatozoa recovered after gradient preparation and at least 3 millions of sperm cells in the ejaculate
* First Assisted reproductive technology (ART) attempt

Exclusion Criteria:

* Female age > 38
* Female follicle stimulating hormone (FSH) level > 9

Ages: 18 Years to 38 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 255 (Actual)
Dates: Start 2008-10; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Number of Delivery | 9 months

SECONDARY OUTCOMES:
Implantation rate | 3 months
  Number of fetal heart beat/ number of transferred embryos

CONTACTS AND LOCATIONS:
Overall Officials: Jean PARINAUD, MD, PhD, Study Chair — University Hospital, Toulouse
Locations (9):
- France (9):
  - Bagnolet Hospital, Bagnolet
  - Laboratoire CLEMENT, Le Blanc-Mesnil
  - Laboratoire de Biologie de la Reproduction, Hôpital Jeanne de Flandre, Lille
  - Institut Mutualiste Montsouris, Paris
  - Hôpital Bichat, Paris
  - Service de génétique et Biologie de la Reproduction CECOS, Hôpital Maison Blanche, Reims
  - Laboratoire de Biologie de la Reproduction CECOS, Rouen
  - Cmco-Sihcus, Schiltigheim
  - CH des 4 villes, Sèvres